CLINICAL TRIAL: NCT02499770
Title: Phase 1b/2a Safety and Pharmacokinetic Study of G1T28 in Patients With Extensive Stage Small Cell Lung Cancer (SCLC) Receiving Etoposide and Carboplatin
Brief Title: Trilaciclib (G1T28), a CDK 4/6 Inhibitor, in Combination With Etoposide and Carboplatin in Extensive Stage Small Cell Lung Cancer (SCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G1T28-02; 2016-001583-11 (EudraCT Number)
Record Dates: First submitted 2015-07-08; First posted 2015-07-16 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; CDK 4/6 Inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; trilaciclib; Etoposide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- trilaciclib + carboplatin/etoposide (Experimental): All patients in part 1 will receive trilaciclib (G1T28) prior to standard chemotherapy- carboplatin and etoposide. Patients will have PK assessments completed on days 1 and 3 in cycle 1 only. All patents will be monitored for safety and tumor response based on RECIST version 1.1. Safety surveillance reporting of AEs and concomitant medications commences at the time that informed consent is obtained and continues through the Post Treatment Visit.
  Interventions: Drug: Carboplatin; Drug: Trilaciclib; Drug: Etoposide
- trilaciclib/placebo + carboplatin/etoposide (Experimental): All patients enrolled in part 2 will be randomized to receive either trilaciclib (G1T28) or placebo administered prior to standard chemotherapy- carboplatin and etoposide. All patents will be monitored for safety and tumor response based on RECIST version 1.1. Safety surveillance reporting of AEs and concomitant medications commences at the time that informed consent is obtained and continues through the Post Treatment Visit.
  Interventions: Drug: Carboplatin; Drug: Placebo; Drug: Trilaciclib; Drug: Etoposide

INTERVENTIONS:
Drug: Carboplatin
  Other Names: Paraplatin
Drug: Placebo
  Arms: trilaciclib/placebo + carboplatin/etoposide
Drug: Trilaciclib
  Other Names: G1T28
Drug: Etoposide
  Other Names: VP-16; Toposar

SUMMARY:
This is a study to investigate the potential clinical benefit of trilaciclib (G1T28) in preserving the bone marrow and the immune system, and enhancing chemotherapy antitumor efficacy when administered prior to carboplatin and etoposide in first line treatment for patients with newly diagnosed extensive-stage SCLC.

The study consists of 2 parts: a limited open-label, dose-finding portion (Part 1), and a randomized double-blind portion (Part 2). Both parts include 3 study phases: Screening Phase, Treatment Phase, and Survival Follow-up Phase. The Treatment Phase begins on the day of first dose with study treatment and completes at the Post-Treatment Visit. Approximately, 90 patients will be enrolled in the study; 20 patients in the Part 1 and 70 patients in the Part 2 portion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 years
* Unequivocally confirmed diagnosis of SCLC by histology or cytology, preferably including the presence of neuroendocrine features by immunohistochemistry
* At least 1 target lesion that is unirradiated and measurable by RECIST, Version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Adequate organ function

Exclusion Criteria:

* Prior chemotherapy for extensive-stage SCLC
* Presence of symptomatic brain metastases requiring immediate treatment with radiation therapy or steroids.
* Uncontrolled ischemic heart disease or uncontrolled symptomatic congestive heart failure
* Known history of stroke or cerebrovascular accident within 6 months prior to enrollment
* Other uncontrolled serious chronic disease or conditions that in the investigator's opinion could affect compliance or follow-up in the protocol
* Concurrent radiotherapy to any site or radiotherapy within 2 weeks prior to enrollment or previous radiotherapy to the target lesion sites (the sites that are to be followed for determination of a response)
* Receipt of any investigational medication within 4 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2019-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Contact, Study Director — G1 Therapeutics, Inc.
Locations (40):
- United States (26):
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Memorial Hospital - Univ. of Colorado Health, Colorado Springs, Colorado
  - University of Colorado Health, Oncology Clinical Research Northern Region, Fort Collins, Colorado
  - Boca Raton Regional Hospital - Lynn Cancer Institute, Boca Raton, Florida
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists - North, Tavares, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - University Cancer and Blood Center, LLC, Athens, Georgia
  - Emory University, Atlanta, Georgia
  - Norton Cancer Institute, Louisville, Kentucky
  - Center For Cancer and Blood Disorders, Bethesda, Maryland
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Roswell Park, Buffalo, New York
  - UNC - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Oklahoma University - Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Gibbs Cancer Center, Spartanburg, South Carolina
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Hanna Cancer Associates - University of Tennessee, Knoxville, Tennessee
  - Texas Oncology, Tyler, Texas
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
- CHU de Rennes Hopital Pontchaillou, Rennes, France
- ARENSIA Exploratory Medicine LLC, Tbilisi, Georgia
- Hungary (3):
  - Veszprem Megyei Tudogyogyintezet, Farkasgyepű, Veszprém megye
  - Orszagos Koranyi Tbc es Pulmonologiai Intezet, XI. Tudobelosztaly, Budapest
  - Hetenyi Geza Korhaz, Szolnok
- ARENSIA Exploratory Medicine Phase I Unit, The Institute of Oncology, Chisinau, Moldova
- Poland (3):
  - Samodzielny Publiczny ZespAA GruAicy i ChorAb PA¿uc, Olsztyn
  - Wojewodzki Szpital Zespolony im. L. Rydygiera, Torun
  - Centrum Onkologii-Instytut im. Marii Sklodowskiej-Curie, Warsaw
- Spain (5):
  - Hospital Regional Universitario HRU Carlos Haya Malaga, Málaga, Andalusia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Consorcio Hospitalario Provincial, Castillón
  - Hgu Gregorio Maranon, Madrid
  - Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hussein M, Maglakelidze M, Richards DA, Sabatini M, Gersten TA, Lerro K, Sinielnikov I, Spira A, Pritchett Y, Antal JM, Malik R, Beck JT. Myeloprotective Effects of Trilaciclib Among Patients with Small Cell Lung Cancer at Increased Risk of Chemotherapy-Induced Myelosuppression: Pooled Results from Three Phase 2, Randomized, Double-Blind, Placebo-Controlled Studies. Cancer Manag Res. 2021 Aug 9;13:6207-6218. doi: 10.2147/CMAR.S313045. eCollection 2021. PMID 34408488
- [Derived] Ferrarotto R, Anderson I, Medgyasszay B, Garcia-Campelo MR, Edenfield W, Feinstein TM, Johnson JM, Kalmadi S, Lammers PE, Sanchez-Hernandez A, Pritchett Y, Morris SR, Malik RK, Csoszi T. Trilaciclib prior to chemotherapy reduces the usage of supportive care interventions for chemotherapy-induced myelosuppression in patients with small cell lung cancer: Pooled analysis of three randomized phase 2 trials. Cancer Med. 2021 Sep;10(17):5748-5756. doi: 10.1002/cam4.4089. Epub 2021 Aug 18. PMID 34405547
- [Derived] Li C, Hart L, Owonikoko TK, Aljumaily R, Rocha Lima CM, Conkling PR, Webb RT, Jotte RM, Schuster S, Edenfield WJ, Smith DA, Sale M, Roberts PJ, Malik RK, Sorrentino JA. Trilaciclib dose selection: an integrated pharmacokinetic and pharmacodynamic analysis of preclinical data and Phase Ib/IIa studies in patients with extensive-stage small cell lung cancer. Cancer Chemother Pharmacol. 2021 May;87(5):689-700. doi: 10.1007/s00280-021-04239-9. Epub 2021 Feb 17. PMID 33595690
- [Derived] Lai AY, Sorrentino JA, Dragnev KH, Weiss JM, Owonikoko TK, Rytlewski JA, Hood J, Yang Z, Malik RK, Strum JC, Roberts PJ. CDK4/6 inhibition enhances antitumor efficacy of chemotherapy and immune checkpoint inhibitor combinations in preclinical models and enhances T-cell activation in patients with SCLC receiving chemotherapy. J Immunother Cancer. 2020 Oct;8(2):e000847. doi: 10.1136/jitc-2020-000847. PMID 33004541
- [Derived] Weiss JM, Csoszi T, Maglakelidze M, Hoyer RJ, Beck JT, Domine Gomez M, Lowczak A, Aljumaily R, Rocha Lima CM, Boccia RV, Hanna W, Nikolinakos P, Chiu VK, Owonikoko TK, Schuster SR, Hussein MA, Richards DA, Sawrycki P, Bulat I, Hamm JT, Hart LL, Adler S, Antal JM, Lai AY, Sorrentino JA, Yang Z, Malik RK, Morris SR, Roberts PJ, Dragnev KH; G1T28-02 Study Group. Myelopreservation with the CDK4/6 inhibitor trilaciclib in patients with small-cell lung cancer receiving first-line chemotherapy: a phase Ib/randomized phase II trial. Ann Oncol. 2019 Oct 1;30(10):1613-1621. doi: 10.1093/annonc/mdz278. PMID 31504118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 71 centers in the United States of America and Europe. The first participant enrolled on 26 June 2015 and the last participant completed on 22 February 2019. For Part 1, participants were enrolled from 26 June 2015 to 30 September 2016 and for Part 2, participants were enrolled from 06 October 2016 to 25 April 2017.
Pre-assignment Details: Participants were screened within 14 days prior to first study drug administration. Informed consent and brain scans were obtained up to 28 days prior to first study drug administration. A total of 122 participants were enrolled (24 in Part 1 and 98 in Part 2), of which 96 were assigned to treatment.
Groups:
- Part 1: Dose Finding/Expansion: The 1st cohort in Part 1 received trilaciclib 200 mg/m^2, IV once daily on Days 1 to 3 of each 21-day E/P cycle. The 2nd cohort in the Phase 1b dose-finding portion of Part 1 & the Phase 2a expansion cohort in Part 1 received trilaciclib 240 mg/m^2, IV once daily on Days 1 to 3 of each 21-day E/P cycle. Participants received standard E/P chemotherapy in 21-day cycles. Carboplatin dose was calculated using the Calvert formula with a target AUC = 5 (maximum 750 mg) IV on Day 1. Etoposide 100 mg/m^2 was given IV daily on Days 1, 2, & 3 of each 21-day cycle. Trilaciclib was only given with E/P therapy. If E/P therapy was discontinued, trilaciclib was also to be discontinued. The interval between doses of trilaciclib on successive days was not greater than 28 hours & between the dose of trilaciclib & the first dose of chemotherapy on a given day (etoposide or carboplatin) not greater than 4 hours.
- Part 2: Trilaciclib/Placebo IV With E/P: Eligible participants were randomized (1:1) to trilaciclib or placebo administered IV once daily on Days 1 to 3 with etoposide and carboplatin on Day 1 and etoposide on Days 2 and 3 of 21-day cycles (E/P). Randomization was stratified by ECOG performance status (0 to 1 versus 2). Participants received trilaciclib 240 mg/m^2 (recommended dose from Part 1) or placebo IV once daily on Days 1 to 3 of each 21-day E/P chemotherapy cycle. Participants received standard E/P chemotherapy in 21-day cycles. The carboplatin dose was calculated using the Calvert formula with a target AUC = 5 (maximum 750 mg) IV on Day 1, and 100 mg/m^2 etoposide was administered IV daily on Days 1, 2, and 3 of each 21-day cycle. The interval between doses of trilaciclib/placebo on successive days was not greater than 28 hours and between the dose of trilaciclib/placebo and the first dose of chemotherapy on a given day (etoposide or carboplatin) was not greater than 4 hours.
Period: Overall Study
Arm/Group | Part 1: Dose Finding/Expansion | Part 2: Trilaciclib/Placebo IV With E/P
Started | 19 | 77
Completed | 0 | 0
Not Completed | 19 | 77
Not completed — Death | 17 | 56
Not completed — Study completion | 1 | 10
Not completed — Withdrawal by Subject | 0 | 7
Not completed — Lost to Follow-up | 0 | 2
Not completed — Subject declined further treatment | 1 | 0
Not completed — Withdrawn by PI for compassionate reason | 0 | 1
Not completed — Randomized but not enrolled | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants randomized
Groups:
- Part 2: Trilaciclib/Placebo IV With E/P: Eligible participants were randomized (1:1) to trilaciclib or placebo administered IV once daily on Days 1 to 3 of E/P therapy. Randomization was stratified by ECOG performance status (0 to 1 versus 2). Participants received trilaciclib 240 mg/m^2 (recommended dose from Part 1) or placebo IV once daily on Days 1 to 3 of each 21-day E/P chemotherapy cycle. Participants received standard E/P chemotherapy in 21-day cycles. The carboplatin dose was calculated using the Calvert formula with a target AUC = 5 (maximum 750 mg) IV on Day 1, and 100 mg/m^2 etoposide was administered IV daily on Days 1, 2, and 3 of each 21-day cycle. The interval between doses of trilaciclib/placebo on successive days was not greater than 28 hours and between the dose of trilaciclib/placebo and the first dose of chemotherapy on a given day (etoposide or carboplatin) was not greater than 4 hours.
- Total: Total of all reporting groups
Arm/Group | Part 1: Dose Finding/Expansion | Part 2: Trilaciclib/Placebo IV With E/P | Total
Number analyzed (Participants) | 19 | 77 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 37 | 44
  >=65 years | 12 | 40 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 23 | 31
  Male | 11 | 54 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 18 | 75 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 16 | 73 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Country [Count of Participants; unit: Participants]
  United States | 19 | 39 | 58
  Non-United States | 0 | 38 | 38
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Population: BSA was only available for 75 of the 77 participants in Part 2.
  m^2
    number analyzed (Participants) | 19 | 75 | 94
    (all) | 1.90 (0.263) | 1.90 (0.216) | NA (NA) — Mean body surface area was not calculated for all participants overall.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities by Cohort in Cycle 1, Part 1
Description: Dose-limiting toxicities (DLTs) were drug-related toxicities defined as follows:
  1. Absolute neutrophil count (ANC) < 0.5 × 10^9/L lasting for ≥ 7 days
  2. ≥ Grade 3 neutropenic infection/febrile neutropenia
  3. Grade 4 thrombocytopenia (TCP) or ≥ Grade 3 TCP with bleeding
  4. Unable to start next cycle of chemotherapy due to lack of recovery to an ANC ≥ 1.5 × 10^9/L and platelet count ≥ 100 × 10^9/L
  5. ≥ Grade 3 nonhematologic toxicity (nausea, vomiting, and diarrhea failing maximal medical management; fatigue lasting for > 72 hours)
  Toxicities not clearly related to etoposide/carboplatin therapy were also considered for the purposes of determining DLTs.
Time Frame: Days 1-21 of Cycle 1
Population: Safety analysis set - included all enrolled participants (i.e., signed informed consent) who received at least 1 dose of study drug (etoposide, carboplatin, or trilaciclib).
  Part 1: Cohort 1 Trilaciclib 200 mg/m^2 included 1 participant from Part 2 and 1 participant from Part 1 240 mg/m^2 who received 200 mg/m^2.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Cohort 1 Trilaciclib 200 mg/m^2: Participants received trilaciclib 200 mg/m^2 administered intravenously (IV) once daily on Days 1 to 3 of each 21-day E/P chemotherapy cycle.
- Part 1: Cohort 2 Trilaciclib 240mg/m^2: Participants received trilaciclib 240 mg/m^2 administered IV once daily on Days 1 to 3 of each 21-day E/P chemotherapy cycle.
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 12 | 8
Participants
  Number of participants meeting ≥1 DLT criteria | 2 | 1
  Grade 4 TCP or ≥Grade 3 TCP with bleeding | 1 | 0
  Unable to start next cycle of chemotherapy | 1 | 1

2. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Related AEs, Related SAEs, and AEs Leading to Study Drug Discontinuation in Part 1
Description: An AE was defined as any untoward medical occurrence in a participant administered a medicinal product that did not necessarily have a causal relationship with this treatment. TEAEs were defined as any AE that started on or after the first dose of study drug and up to the last dose +30 days. SAEs were defined as any untoward medical occurrence that at any dose resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or was a congenital anomaly/birth defect. Relatedness to study drug was assessed by the investigator. Related refers to those events that were Possibly, Probably, or Definitely Related. AEs with an unknown/not reported onset date were also included.
Time Frame: TEAEs were any AE that started on or after the first dose of study drug and up to the last dose +30 days (a minimum of 51 days up to a maximum of 374 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 12 | 8
Participants
  Any TEAE | 12 | 8
  Any SAE | 4 | 1
  TEAE related to any study drug | 10 | 8
  SAE related to any study drug | 0 | 0
  TEAE leading to discontinuation of any study drug | 0 | 0

3. Primary Outcome: Duration of Severe (Grade 4) Neutropenia in Part 2
Description: Severe (Grade 4) neutropenia was defined as at least 1 ANC value <0.5 × 10^9/L during the treatment period. Within each cycle, the duration (days) of severe neutropenia was defined as the number of days from the date of the first ANC value of <0.5 × 10^9/L observed between start of cycle and end of cycle to the date of the first ANC value ≥0.5 × 10^9/L that met the following criteria: 1) occurred after the ANC value of <0.5 × 10^9/L and 2) no other ANC values <0.5 × 10^9/L occurred between this day and end of cycle. The duration of severe neutropenia only included participants who had at least 1 severe neutropenia event in the cycle, and censoring rules were applied for unresolved severe neutropenia in a cycle. For the treatment period, the overall duration of severe neutropenia was the median value among the durations from all cycles.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: Full analysis set (FAS) - included all randomized participants who received at least 1 dose of study drug (etoposide, carboplatin, or trilaciclib). Analyses using the FAS were conducted on the basis of the assigned treatment.
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Part 2: Placebo: Participants received placebo IV once daily on Days 1 to 3 of each 21-day E/P chemotherapy cycle.
- Part 2: Trilaciclib 240 mg/m^2: Participants received trilaciclib 240 mg/m^2 IV once daily on Days 1 to 3 of each 21-day E/P chemotherapy cycle.
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 16 | 2
Days | 8 [7 to 8] | 3 [2 to 3]
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: Trilaciclib 240 mg/m^2; Test type: Other; p = 0.0097, Stratified log-rank test — The p-value was calculated using the stratified log-rank test to account for the baseline ECOG status (0-1 vs 2) as the stratification factor. Significance level was set as two-sided 0.2; p-value calculated using stratified log-rank test with baseline ECOG status (0-1 vs 2) as stratification factor. Significance level was two-sided 0.2

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Trilaciclib in Cycle 1, Part 1
Description: Cmax of trilaciclib in plasma was determined from individual concentration-time data by non-compartmental analysis methods. The actual sampling times in relation to dosing were used. For estimation of Cmax, a concentration that was below the limit of quantification (BLQ) was assigned a value of zero if it occurred in a profile before the first measurable concentration. If a BLQ value occurred after a measurable concentration in a profile, and was followed by a value above the lower limit of quantification, then the BLQ was treated as missing data. If a BLQ value occurred at the end of the collection interval (after the last quantifiable concentration) it was treated as missing data. If two BLQ values occurred in succession after Cmax, the profile was deemed to have terminated at the first BLQ value and any subsequent concentrations were omitted.
Time Frame: Days 1 and 3 of Cycle 1 for a 21-day cycle
Population: Pharmacokinetic (PK) analysis set - included all participants with evaluable PK profiles for both treatments and analytes.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 8 | 1
ng/mL
  Day 1 Cycle 1 | 1240 (738) | 1570 (NA) — Not calculable
  Day 3 Cycle 1 | 1620 (1040) | 2260 (NA) — Not calculable

5. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) for Trilaciclib in Cycle 1, Part 1
Description: AUC0-inf of trilaciclib in plasma was determined from individual concentration-time data by non-compartmental analysis methods. The actual sampling times in relation to dosing were used.
Time Frame: Days 1 and 3 of Cycle 1 for a 21-day cycle
Population: PK analysis set - included all participants with evaluable PK profiles for both treatments and analytes
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 8 | 1
h*ng/mL
  Day 1 Cycle 1 | 2560 (792) | 2280 (NA) — Not calculable (n=1)
  Day 3 Cycle 1 | 3110 (693) | 2960 (NA) — Not calculable (n=1)

6. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of Trilaciclib in Cycle 1, Part 1
Description: Tmax of trilaciclib in plasma was determined from individual concentration-time data by non-compartmental analysis methods. The actual sampling times in relation to dosing were used.
Time Frame: Days 1 and 3 of Cycle 1 for a 21-day cycle
Population: PK analysis set - included all participants with evaluable PK profiles for both treatments and analytes
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 8 | 1
Hours
  Day 1 Cycle 1 | 0.57 [0.45 to 0.98] | 0.50 [NA to NA] — Not calculable (n=1)
  Day 3 Cycle 1 | 0.52 [0.47 to 1.00] | 0.45 [NA to NA] — Not calculable (n=1)

7. Secondary Outcome: Cmax of Etoposide and Free and Total Carboplatin in Cycle 1, Part 1
Description: Cmax of etoposide and free and total carboplatin in plasma were determined from individual concentration-time data by non-compartmental analysis methods. The actual sampling times in relation to dosing were used. For estimation of Cmax, a concentration that was BLQ was assigned a value of zero if it occurred in a profile before the first measurable concentration. If a BLQ value occurred after a measurable concentration in a profile, and was followed by a value above the lower limit of quantification, then the BLQ was treated as missing data. If a BLQ value occurred at the end of the collection interval (after the last quantifiable concentration) it was treated as missing data. If two BLQ values occurred in succession after Cmax, the profile was deemed to have terminated at the first BLQ value and any subsequent concentrations were omitted.
Time Frame: Days 1 and 3 of Cycle 1 for a 21-day cycle (carboplatin was only dosed on Day 1 so there are no Day 3 Cmax values)
Population: PK analysis set - included all participants with evaluable PK profiles for both treatments and analytes
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part 1: Dose Finding/Expansion
Number analyzed (Participants) | 9
μg/mL
  Etoposide Day 1 Cycle 1 | 21.9 (2.70)
  Etoposide Day 3 Cycle 1 | 20.2 (2.40)
  Free Carboplatin Day 1 Cycle 1 | 20.3 (6.83)
  Total Carboplatin Day 1 Cycle 1 | 18.8 (5.45)

8. Secondary Outcome: AUC0-inf of Etoposide and Free and Total Carboplatin in Cycle 1, Part 1
Description: AUC0-inf of etoposide and free and total carboplatin in plasma were determined from individual concentration-time data by non-compartmental analysis methods. The actual sampling times in relation to dosing were used.
Time Frame: Days 1 and 3 of Cycle 1 for a 21-day cycle (carboplatin was only dosed on Day 1 so there are no Day 3 AUC0-inf values)
Population: PK analysis set - included all participants with evaluable PK profiles for both treatments and analytes
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Part 1: Dose Finding/Expansion
Number analyzed (Participants) | 9
h*μg/mL
  Etoposide Day 1 Cycle 1: number analyzed (Participants) | 8
  Etoposide Day 1 Cycle 1 | 131 (44.7)
  Etoposide Day 3 Cycle 1 | 146 (48.4)
  Free Carboplatin Day 1 Cycle 1: number analyzed (Participants) | 7
  Free Carboplatin Day 1 Cycle 1 | 50.5 (14.4)
  Total Carboplatin Day 1 Cycle 1 | 137 (37.3)

9. Secondary Outcome: Tmax of Etoposide and Free and Total Carboplatin in Cycle 1, Part 1
Description: Tmax of etoposide and free and total carboplatin in plasma was determined from individual concentration-time data by non-compartmental analysis methods. The actual sampling times in relation to dosing were used.
Time Frame: Days 1 and 3 of Cycle 1 for a 21-day cycle (carboplatin was only dosed on Day 1 so there are no Day 3 Tmax values)
Population: PK analysis set - included all participants with evaluable PK profiles for both treatments and analytes
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Dose Finding/Expansion
Number analyzed (Participants) | 9
Hours
  Etoposide Day 1 Cycle 1 | 1.08 [0.90 to 2.67]
  Etoposide Day 3 Cycle 1 | 1.00 [0.85 to 1.52]
  Free Carboplatin Day 1 Cycle 1 | 0.52 [0.47 to 0.67]
  Total Carboplatin Day 1 Cycle 1 | 0.52 [0.47 to 0.67]

10. Secondary Outcome: Duration of Severe (Grade 4) Neutropenia in Part 1
Description: as for outcome 3
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: The FAS included all randomized patients who received at least 1 dose of study drug (etoposide, carboplatin, or trilaciclib). Analyses using the FAS were conducted on the basis of the assigned treatment. No participants had severe (Grade 4) neutropenia in the 240 mg/m^2 arm.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 4 | 0
Days | 6 [6 to 7] |

11. Secondary Outcome: Occurrence of Severe (Grade 4) Neutropenia in Part 1
Description: Severe (Grade 4) neutropenia was defined as at least 1 ANC value <0.5 × 10^9/L during the treatment period.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: The FAS included all randomized patients who received at least 1 dose of study drug (etoposide, carboplatin, or trilaciclib). Analyses using the FAS were conducted on the basis of the assigned treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Participants | 4 | 0

12. Secondary Outcome: Occurrence of Febrile Neutropenia in Part 1
Description: Each febrile neutropenia event (as defined by Common Terminology Criteria for Adverse Events [CTCAE]) was captured as an AE. The occurrence of febrile neutropenia was defined as at least 1 febrile neutropenia event during the treatment period. For the treatment period, the total number of febrile neutropenia events was the number of febrile neutropenia events with a unique start date.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

13. Secondary Outcome: Duration of Grade 3/4 Neutropenia in Part 1
Description: Grade 3/4 neutropenia was defined as at least 1 ANC value <1.0 × 10^9/L during the treatment period. Within each cycle, duration (days) of Grade 3/4 neutropenia was defined as the number of days from the date of the first ANC value of <1.0 × 10^9/L observed between start of cycle and end of cycle to the date of the first ANC value ≥1.0 × 10^9/L that met the following criteria: 1) occurred after the ANC value of <1.0 × 10^9/L and 2) no other ANC values <1.0 × 10^9/L occurred between this day and end of cycle. The duration of Grade 3/4 neutropenia only included participants who had at least 1 Grade 3/4 neutropenia event in the cycle, and censoring rules were applied for unresolved Grade 3/4 neutropenia in a cycle. For the treatment period, the overall duration of Grade 3/4 neutropenia was the median value among the durations of Grade 3/4 neutropenia from all cycles.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 6 | 3
Days | 8 [6 to 10] | 8 [5 to 9]

14. Secondary Outcome: Occurrence of Grade 3/4 Neutropenia in Part 1
Description: Grade 3/4 neutropenia was defined as at least 1 ANC value <1.0 × 10^9/L during the treatment period.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Participants | 6 | 3

15. Secondary Outcome: Nadir of Absolute Neutrophil Count in Cycle 1, Part 1
Description: Cycle nadir was the lowest value for ANC that occurred between start of cycle and end of cycle and was less than the cycle baseline.
Time Frame: From baseline to the end of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: x 10^9 cells/L
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
x 10^9 cells/L | 1.198 (0.7241) | 1.653 (0.7381)

16. Secondary Outcome: Occurrence of Granulocyte-Colony Stimulating Factor (G-CSF) Administration in Part 1
Description: Administration of G-CSF was collected with concomitant medications, which were coded using World Health Organization Drug Dictionary (WHO-DD) Version September 2017. A cycle where G-CSF was administered concurrently was identified by comparing the start and stop dates of each administration of G-CSF to the start of cycle and end of cycle. The occurrence of G-CSF administrations was defined as at least 1 cycle with G-CSF administrations during the treatment period. For the treatment period, the total number of G-CSF administrations was the number of cycles with G-CSF administrations.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Participants | 5 | 3

17. Secondary Outcome: Occurrence of Red Blood Cell (RBC) Transfusion in Part 1
Description: Within a cycle, a RBC transfusion event was defined as either 1) an actual RBC transfusion, or 2) eligible for RBC transfusion (defined as hemoglobin <8.0 g/dL). The occurrence of RBC transfusions was defined as at least 1 cycle with RBC transfusion during the treatment period. For the treatment period, the total number of RBC transfusions was the number of cycles with RBC transfusions.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Participants | 4 | 1

18. Secondary Outcome: Change From Baseline of Hemoglobin at the End of Cycle 6, Part 1
Description: Blood samples were collected for local clinical laboratory assessment of hemoglobin levels.
Time Frame: Baseline, Day 1, Day 3, Day 8, Day 10, and Day 15 of a 21-day cycle x 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 5 | 7
g/L | -9.8 (13.27) | -20.1 (15.21)

19. Secondary Outcome: Occurrence of Erythropoietin Stimulating Agent (ESA) Administration in Part 1
Description: Administration of ESAs was collected with concomitant medications, which were coded using WHO-DD Version September 2017. A cycle where an ESA was administered concurrently was identified by comparing the start and stop dates of each administration of an ESA to the start of cycle and end of cycle. The occurrence of ESA administration was at least 1 cycle with an ESA administration during the treatment period. For the treatment period, the total number of ESA administrations was the number of cycles with ESA administrations.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Participants | 2 | 0

20. Secondary Outcome: Occurrence of Platelet Transfusion in Part 1
Description: Within a cycle, a platelet transfusion event was defined as either 1) an actual platelet transfusion, or 2) eligible for platelet transfusion (defined as a platelet count ≤10 × 10^9/L). The occurrence of platelet transfusions was defined as at least 1 cycle with platelet transfusion during the treatment period. For the treatment period, the total number of platelet transfusions was the number of cycles with platelet transfusions.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Participants | 1 | 0

21. Secondary Outcome: Change From Baseline of Platelet Count at the End of Cycle 6, Part 1
Description: Blood samples were collected for local clinical laboratory assessment of platelet count.
Time Frame: Baseline, Day 1, Day 3, Day 8, Day 10, and Day 15 of a 21-day cycle x 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: x 10^9 cells/L
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 5 | 7
x 10^9 cells/L | -72.6 (88.38) | -59.4 (108.47)

22. Secondary Outcome: Change From Baseline of Lymphocyte Count at the End of Cycle 6, Part 1
Description: Blood samples were collected for local clinical laboratory assessment of lymphocyte count.
Time Frame: Baseline, Day 1, Day 3, Day 8, Day 10, and Day 15 of a 21-day cycle x 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: x 10^9 cells/L
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 5 | 7
x 10^9 cells/L | 0.188 (0.8431) | 0.067 (0.4691)

23. Secondary Outcome: Occurrence of Dose Reduction in Part 1
Description: Dose reductions were not permitted for trilaciclib, per study protocol. Dose reductions for E/P were derived from changes in the protocol-specified dose on the dosing page and corresponded to the reductions for toxicity specified in the protocol. No more than 2 dose reductions of E/P in total were allowed for any participant. Simultaneous reductions in the doses of E/P were counted as 1 dose reduction. For the treatment period, the total number of dose reductions was the number of cycles where there was at least 1 dose reduction.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 12 | 8
Participants | 2 | 3

24. Secondary Outcome: Occurrence of Infectious SAEs in Part 1
Description: SAEs were defined as any untoward medical occurrence that at any dose resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or was a congenital anomaly/birth defect. An infectious SAE was a serious event in the Medical Dictionary for Regulatory Activities (MedDRA) system organ class "infections and infestations" and a preferred term of anal abscess, bacteraemia, bronchitis, candida infection, chronic sinusitis, conjunctivitis, infection, influenza, nasopharyngitis, oral candidiasis, oral herpes, pharyngitis streptococcal, pneumonia, pneumonia bacterial, respiratory tract infection, sepsis, skin infection, upper respiratory tract infection, urinary tract infection, urosepsis or viral upper respiratory tract infection.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Participants | 2 | 1

25. Secondary Outcome: Occurrence of Pulmonary Infection SAE in Part 1
Description: SAEs were defined as any untoward medical occurrence that at any dose resulted in death, was life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or was a congenital anomaly/birth defect. A pulmonary infection SAE was a serious event in the MedDRA system organ class "infections and infestations" and a preferred term of bronchitis, influenza, pneumonia, pneumonia bacterial, respiratory tract infection, upper respiratory tract infection or viral upper respiratory tract infection.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Participants | 1 | 0

26. Secondary Outcome: Occurrence of IV Antibiotic Administration in Part 1
Description: Intravenous antibiotic administration was collected with concomitant medications, which were coded using WHO-DD Version September 2017. A cycle where IV antibiotic was administered concurrently was identified by comparing the start and stop dates of each administration of IV antibiotic to the start of cycle and end of cycle. The occurrence of IV antibiotic administration was defined as at least 1 cycle with IV antibiotic administration during the treatment period. For the treatment period, the total number of IV antibiotic administrations was the number of cycles with IV antibiotic administrations.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Participants | 4 | 1

27. Secondary Outcome: Time to First Major Adverse Hematologic Event (MAHE) in Part 1
Description: MAHE was a composite endpoint incorporating the measurement of several clinically meaningful aspects of myelopreservation into a single endpoint. The individual components for MAHE were hospitalization for a hematologic event, febrile neutropenia, death related to treatment, dose delay/reduction due to ANC or platelet counts, prolonged severe neutropenia (duration >5 days), RBC transfusion (actual or eligible) and platelet transfusion (actual or eligible). Time to first occurrence of a MAHE event was defined as the first time to observe an interested event among all the components, starting from the first dose date of study drug administration.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Months | 2.6 [0.8 to NA] — Not evaluable | 3.0 [1.0 to NA] — Not evaluable

28. Secondary Outcome: Best Overall Tumor Response Based on Assessments in Part 1
Description: Tumor response was assessed by computed tomography (CT) or magnetic resonance imaging (MRI). Overall visit response by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 was derived programmatically using data from target lesions (TLs), non-target lesions (NTLs), & new lesions. Tumor response data were used to determine each participant's time point response & best overall response (BOR). Complete response (CR) was disappearance of all TLs, any pathological lymph nodes selected as TLs must have reduced in short axis to <10 mm. Partial response (PR) was at least a 30% decrease from baseline in the sum of diameters of TLs, as long as criteria for progressive disease (PD) were not met. PD was a ≥20% increase in the smallest sum of diameters of TLs since treatment started (including baseline) and an absolute increase of ≥5 mm. Stable disease (SD) was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Baseline, end of every two 21-day cycles, up until disease progression to a maximum of the time at least 70% overall survival (OS) events observed (a maximum of 4 years)
Population: Response evaluable analysis set included all participants in the safety analysis set who had at least 1 post-baseline tumor assessment, or clinical progression as noted by the investigator before their first post-baseline tumor scan, or who died due to disease progression before their first post-baseline tumor scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 8
Participants
  CR | 0 | 1
  PR | 8 | 7
  SD | 0 | 0
  PD | 1 | 0
  Not evaluable | 0 | 0
  Unconfirmed CR | 1 | 0
  Unconfirmed PR | 0 | 0

29. Secondary Outcome: Best Overall Tumor Response Based on Blinded Independent Central Review (BICR) Assessments in Part 1
Description: Tumor response was assessed by CT or MRI. Overall visit response by RECIST v1.1 was determined by BICR. Tumor response data were used to determine each participant's time point response & BOR. CR was disappearance of all TLs, any pathological lymph nodes selected as TLs must have reduced in short axis to <10 mm. PR was at least a 30% decrease from baseline in the sum of diameters of TLs, as long as criteria for PD were not met. PD was a ≥20% increase in the smallest sum of diameters of TLs since treatment started (including baseline) and an absolute increase of ≥5 mm. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Baseline, end of every two 21-day cycles, up until disease progression to a maximum of the time at least 70% OS events observed (a maximum of 4 years)
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 8
Participants
  CR | 1 | 0
  PR | 6 | 8
  SD | 2 | 0
  PD | 0 | 0
  Not evaluable | 0 | 0
  Unconfirmed CR | 0 | 0
  Unconfirmed PR | 2 | 0

30. Secondary Outcome: Progression Free Survival (PFS) Based on Assessments in Part 1
Description: Tumor response was assessed by CT or MRI. PFS was defined as the time (months) from date of first dose date of study drug for participants in Part 1 until date of documented disease progression or death due to any cause, whichever occurred first. More specifically, PFS was determined using all the assessment data up until the last evaluable visit prior to or on the date of i) disease progression as defined by RECIST 1.1 or by clinical criteria as determined by the investigator; or ii) withdrawal of consent; or iii) receiving subsequent anticancer therapy, whichever was earlier. For PFS determined using response data derived programmatically, either clinical progression or progression by RECIST (whichever came first) was considered. Median and inter-quartile range of PFS were calculated using the Kaplan-Meier method.
Time Frame: as for outcome 29
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Months | 5.3 [1.5 to 6.1] | 6.3 [5.9 to 9.1]

31. Secondary Outcome: OS in Part 1
Description: OS was calculated as the time (months) from date of first dose of study drug for participants in Part 1 to the date of death due to any cause. Participants who did not die during the study were censored at the date last known to be alive. Participants lacking data beyond the day of first dose of study drug had their survival time censored at day of first dose of study drug. OS was not censored if a participant received other anti-tumor treatments after the study drugs. Median and inter-quartile range of OS were calculated using the Kaplan-Meier method.
Time Frame: Baseline up until death or a maximum of the time at least 70% OS events observed (a maximum of 4 years)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2
Number analyzed (Participants) | 10 | 9
Months | 10.6 [4.9 to 25.1] | 12.8 [9.5 to 13.5]

32. Secondary Outcome: Occurrence of Severe (Grade 4) Neutropenia in Part 2
Description: Severe (Grade 4) neutropenia was defined as at least 1 ANC value <0.5 × 10^9/L during the treatment period.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Participants | 16 | 2

33. Secondary Outcome: Occurrence of Febrile Neutropenia in Part 2
Description: Each febrile neutropenia event (as defined by CTCAE) was captured as an AE. The occurrence of febrile neutropenia was defined as at least 1 febrile neutropenia event during the treatment period. For the treatment period, the total number of febrile neutropenia events was the number of febrile neutropenia events with a unique start date.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Participants | 3 | 1

34. Secondary Outcome: Duration of Grade 3/4 Neutropenia in Part 2
Description: as for outcome 13
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 30 | 14
Days | 8 [7 to 13] | 8 [6 to 8]

35. Secondary Outcome: Occurrence of Grade 3/4 Neutropenia in Part 2
Description: Grade 3/4 neutropenia was defined as at least 1 ANC value <1.0 × 10^9/L during the treatment period.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Participants | 30 | 14

36. Secondary Outcome: Nadir of Absolute Neutrophil Count in Cycle 1, Part 2
Description: as for outcome 15
Time Frame: From baseline to the end of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: x 10^9 cells/L
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 35
x 10^9 cells/L | 0.815 (0.6385) | 1.899 (1.1930)

37. Secondary Outcome: Occurrence of G-CSF Administration in Part 2
Description: Administration of G-CSF was collected with concomitant medications, which were coded using WHO-DD Version September 2017. A cycle where G-CSF was administered concurrently was identified bycomparing the start and stop dates of each administration of G-CSF to the start of cycle and end of cycle. The occurrence of G-CSF administrations was defined as at least 1 cycle with G-CSF administrations during the treatment period. For the treatment period, the total number of G-CSF administrations was the number of cycles with G-CSF administrations.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Participants | 24 | 4

38. Secondary Outcome: Occurrence of RBC Transfusion in Part 2
Description: Within a cycle, a RBC transfusion event was defined as either 1) an actual RBC transfusion, or 2) eligible for RBC transfusion (defined as hemoglobin <8.0 g/dL). The occurrence of RBC transfusions was defined as at least 1 cycle with RBC transfusion during the treatment period. For the treatment period, the total number of RBC transfusions was the number of cycles with RBC transfusions. If a participant did not have any RBC transfusions, they were assigned a value of 0.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Participants
  Overall | 9 | 6
  On/after Week 5 | 9 | 2

39. Secondary Outcome: Change From Baseline of Hemoglobin at the End of Cycle 6, Part 2
Description: Blood samples were collected for local clinical laboratory assessment of hemoglobin levels.
Time Frame: Baseline, Day 1, Day 3, Day 8, Day 10, and Day 15 of a 21-day cycle x 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 22 | 20
g/L | -25.9 (14.63) | -20.6 (13.83)

40. Secondary Outcome: Occurrence of ESA Administration in Part 2
Description: as for outcome 19
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Participants | 2 | 1

41. Secondary Outcome: Occurrence of Platelet Transfusion in Part 2
Description: as for outcome 20
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Participants | 0 | 2

42. Secondary Outcome: Change From Baseline of Platelet Count at the End of Cycle 6, Part 2
Description: Blood samples were collected for local clinical laboratory assessment of platelet count.
Time Frame: Baseline, Day 1, Day 3, Day 8, Day 10, and Day 15 of a 21-day cycle x 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: x 10^9 cells/L
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 22 | 20
x 10^9 cells/L | -32.7 (100.20) | -54.4 (95.44)

43. Secondary Outcome: Change From Baseline of Lymphocyte Count at the End of Cycle 6, Part 2
Description: Blood samples were collected for local clinical laboratory assessment of lymphocyte count.
Time Frame: Baseline, Day 1, Day 3, Day 8, Day 10, and Day 15 of a 21-day cycle x 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: x 10^9 cells/L
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 22 | 20
x 10^9 cells/L | -0.203 (0.4382) | 0.104 (0.6320)

44. Secondary Outcome: Occurrence of Dose Reduction in Part 2
Description: as for outcome 23
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Participants | 13 | 3

45. Secondary Outcome: Occurrence of Infectious SAEs in Part 2
Description: SAEs were defined as any untoward medical occurrence that at any dose resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or was a congenital anomaly/birth defect. An infectious SAE was a serious event in the MedDRA system organ class "infections and infestations" and a preferred term of anal abscess, bacteraemia, bronchitis, candida infection, chronic sinusitis, conjunctivitis, infection, influenza, nasopharyngitis, oral candidiasis, oral herpes, pharyngitis streptococcal, pneumonia, pneumonia bacterial, respiratory tract infection, sepsis, skin infection, upper respiratory tract infection, urinary tract infection, urosepsis or viral upper respiratory tract infection.
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Participants | 2 | 4

46. Secondary Outcome: Occurrence of Pulmonary Infection SAE in Part 2
Description: as for outcome 25
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Trilaciclib 240 mg/m^2: Participants received trilaciclib 240 mg/m^2 IV once daily on Days 1 to 3 of each 21- day E/P chemotherapy cycle.
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Participants | 1 | 4

47. Secondary Outcome: Occurrence of IV Antibiotic Administration in Part 2
Description: as for outcome 26
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Participants | 8 | 8

48. Secondary Outcome: Time to First MAHE in Part 2
Description: as for outcome 27
Time Frame: From randomization to the end of the treatment period (a minimum of 51 days up to a maximum of 379 days)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Months | 1.0 [0.5 to 2.3] | NA [3.3 to NA] — Not evaluable

49. Secondary Outcome: Best Overall Tumor Response Based on Assessments in Part 2
Description: Tumor response was assessed by CT or MRI. Overall visit response by RECIST v1.1 was derived programmatically using data from TLs, NTLs, & new lesions. Tumor response data were used to determine each participant's time point response & BOR. CR was disappearance of all TLs, any pathological lymph nodes selected as TLs must have reduced in short axis to <10 mm. PR was at least a 30% decrease from baseline in the sum of diameters of TLs, as long as criteria for PD were not met. PD was a ≥20% increase in the smallest sum of diameters of TLs since treatment started (including baseline) and an absolute increase of ≥5 mm. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 36
Participants
  CR | 1 | 0
  PR | 19 | 24
  SD | 12 | 9
  PD | 4 | 1
  Not evaluable | 1 | 0
  Unconfirmed CR | 0 | 0
  Unconfirmed PR | 6 | 4

50. Secondary Outcome: Best Overall Tumor Response Based on BICR Assessments in Part 2
Description: as for outcome 29
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 36
Participants
  CR | 0 | 1
  PR | 23 | 23
  SD | 10 | 7
  PD | 4 | 2
  Not evaluable | 0 | 1
  Unconfirmed CR | 0 | 0
  Unconfirmed PR | 5 | 4

51. Secondary Outcome: PFS Based on Assessments in Part 2
Description: as for outcome 30
Time Frame: as for outcome 29
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Months | 5.0 [3.2 to 6.8] | 6.1 [4.2 to 9.5]

52. Secondary Outcome: OS in Part 2
Description: OS was calculated as the time (months) from date of first dose of study drug for participants in Part 2 to the date of death due to any cause. Participants who did not die during the study were censored at the date last known to be alive. Participants lacking data beyond the day of first dose of study drug had their survival time censored at day of first dose of study drug. OS was not censored if a participant received other anti-tumor treatments after the study drugs. Median and inter-quartile range of OS were calculated using the Kaplan-Meier method.
Time Frame: Baseline up until death or a maximum of the time at least 70% OS events observed (a maximum of 4 years)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 38
Months | 10.6 [6.9 to 16.9] | 10.9 [7.3 to 20.1]

53. Post Hoc Outcome: Duration of Severe (Grade 4) Neutropenia in Cycle 1 of Part 2
Description: In addition to deriving severe (Grade 4) neutropenia using the method described for the primary endpoints, an approach was applied that accounted for participants who did not experience a severe neutropenia event in Cycle 1. For the post-hoc analysis, severe neutropenia was defined as at least 1 ANC value <0.5 × 10^9/L during the treatment period. In Cycle 1, the duration (days) of severe neutropenia was defined as the number of days from the date of the first ANC value of <0.5 × 10^9/L observed between start of cycle and end of cycle to the date of the first ANC value ≥0.5 × 10^9/L that met the following criteria: 1) occurred after the ANC value of <0.5 × 10^9/L and 2) no other ANC values <0.5 × 10^9/L occurred between this day and end of cycle. The duration of severe neutropenia was set to 0 for participants who did not experience severe neutropenia in Cycle 1. Data from unscheduled visits and the actual assessment date (rather than visit date) were included in the derivation.
Time Frame: From baseline to the end of Cycle 1
Population: as for outcome 11
Measure: Median (Full Range); unit: Days
Arm/Group | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
Number analyzed (Participants) | 37 | 36
Days | 0 [0 to 13] | 0 [0 to 3]

ADVERSE EVENTS:
Time Frame: All AEs occurring from the first date of administration of trilaciclib or placebo + E/P therapy through and including 30 calendar days after the last administration of trilaciclib or placebo + E/P therapy were recorded (a minimum of 51 days up to a maximum of 374 days).
Description: AEs are reported for the safety analysis set which included all enrolled participants (i.e., signed informed consent) who received at least 1 dose of study drug (etoposide, carboplatin, or trilaciclib). Analyses using the safety analysis set were conducted on the basis of the actual treatment.
Groups:
- Part 1: Cohort 1 Trilaciclib 200 mg/m^2: Participants received trilaciclib 200 mg/m^2 administered intravenously (IV) once daily on Days 1 to 3 of each 21-day E/P chemotherapy cycle. One participant was screened and dosed at trilaciclib 200 mg/m^2 for Part 2 of the study without being randomized. AEs for this participant are summarized under the Part 1 trilaciclib 200 mg/m^2 cohort for the safety analysis set. One participant was enrolled in the Part 1 trilaciclib 240 mg/m^2 cohort, but dosed at trilaciclib 200 mg/m^2. AEs for this participant's are presented in the trilaciclib 200 mg/m^2 cohort for the safety analysis set.
Arm/Group | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 | Part 1: Cohort 2 Trilaciclib 240mg/m^2 | Part 2: Placebo | Part 2: Trilaciclib 240 mg/m^2
All-Cause Mortality (participants affected / at risk) | 9/12 | 8/8 | 28/37 | 28/38
Serious Adverse Events (participants affected / at risk) | 4/12 | 1/8 | 9/37 | 11/38
Other Adverse Events (participants affected / at risk) | 12/12 | 8/8 | 36/37 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 (N=12) | Part 1: Cohort 2 Trilaciclib 240mg/m^2 (N=8) | Part 2: Placebo (N=37) | Part 2: Trilaciclib 240 mg/m^2 (N=38)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Anemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea hemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Cohort 1 Trilaciclib 200 mg/m^2 (N=12) | Part 1: Cohort 2 Trilaciclib 240mg/m^2 (N=8) | Part 2: Placebo (N=37) | Part 2: Trilaciclib 240 mg/m^2 (N=38)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 3 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (3) | 9 (32) | 3 (9)
Blood creatinine increased (Investigations) | 1 (4) | 2 (3) | 1 (1) | 2 (3)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 4 (12) | 3 (11)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 5 (5) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (5) | 5 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 5 (30) | 5 (14) | 23 (76) | 9 (17)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (18) | 2 (8) | 10 (35) | 10 (12)
Anemia (Blood and lymphatic system disorders) | 5 (21) | 1 (3) | 15 (45) | 10 (19)
Leukopenia (Blood and lymphatic system disorders) | 5 (29) | 0 (0) | 5 (13) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 3 (5) | 5 (5) | 4 (5)
Headache (Nervous system disorders) | 4 (12) | 0 (0) | 3 (4) | 7 (7)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Fatigue (General disorders) | 7 (12) | 4 (10) | 6 (6) | 16 (21)
Edema peripheral (General disorders) | 2 (3) | 2 (4) | 2 (2) | 3 (4)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (5)
Asthenia (General disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 3 (5) | 1 (1) | 5 (5) | 1 (1)
Chills (General disorders) | 2 (5) | 0 (0) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (13) | 4 (8) | 8 (9) | 13 (16)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (5) | 8 (8) | 9 (14)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 2 (3) | 7 (10) | 6 (11)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (13)
Vomiting (Gastrointestinal disorders) | 4 (7) | 4 (7) | 5 (5) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (4) | 11 (14) | 6 (6)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 3 (5) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (7) | 3 (5) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 2 (2) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (4) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (7) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (2) | 2 (2) | 2 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 2 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator will submit results communications for review by the sponsor at least 60 days prior to expected submission to the intended publisher or meeting committee. This review period may be shortened upon mutual consent. The sponsor may request modification of any publication, presentation or use by the investigator if such activity may jeopardize a patent application, an existing patent, or other proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT02499770/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT02499770/SAP_001.pdf